CLINICAL TRIAL: NCT05992519
Title: Diagnostic and Translational Values of Point-of-care Blood Eosinophils and Exhaled Nitric Oxide (FeNO) in People Referred by Primary Care for Suspected Asthma (DIVE)
Brief Title: Diagnostic and Translational Values of Point-of-care Blood Eosinophils and Exhaled Nitric Oxide (FeNO) in People Referred by Primary Care for Suspected Asthma
Acronym: DIVE
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Association Pulmonaire du Quebec (Other); Réseau de Recherche en Santé Respiratoire du Québec (Unknown); AstraZeneca (Industry); Fonds de la Recherche en Santé du Québec (Other Government); Fondation JA DeSève (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-4791
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Asthma; Asthma in Children; Diagnosis; Inflammation
MeSH Terms: conditions — Asthma; Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, whole blood
  Nasosorption for NELF (nasal epithelial lining fluid)
  Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People suspected with asthma: Patients will receive an in invitation letter at the time of BPT scheduling. In the week proceeding the test, the clinical inhalation therapist will discuss the project and schedule the study visit on the day of the BPT. The study visit will be done prior to BPT whenever possible.
  Baseline visit:
  * Medical history
  * 5-item Asthma Control Questionnaire (ACQ-5)
  * FeNO measurement (NIOX VERO device)
  * Nasosorption for nasal epithelial lining fluid (NELF) biobanking
  * blood tests (complete blood count with differential, C-reactive protein, total and specific serum immunoglobulin E, biobank)
  * urine sample (biobank)
  Interventions: Diagnostic Test: ¸FeNO

INTERVENTIONS:
Diagnostic Test: ¸FeNO — FeNO measured with a NIOX VERO device after the methacholine challenge

SUMMARY:
Asthma is characterised by episodic symptoms (attacks) caused by airway inflammation and decreased airflow to the lungs. It affects 10% of the Canadian population and is the most common chronic disease in childhood. Despite its burden and its potential to be life-threatening, establishing the diagnosis takes time due to difficulty in accessing specialised breathing tests. Indeed, the current diagnostic strategy relies on a breathing test (spirometry) and, if non-diagnostic, a subsequent more complicated breathing test conducted in hospitals (a bronchial provocation test). Our dependence on the latter test must be confronted to the bottleneck created by our reliance on it and the difficulty to do these tests in children. Furthermore, within the current framework, people receiving a diagnosis do not know if they have active airway inflammation - a key feature with predicts increased susceptibility to asthma attacks and treatment responsiveness.

Our study's goal is to validate clinically accessible and useful diagnostic tests for peoplesuspected to have asthma. Specifically, we are interested in alternative tests that are a) achievable outside the hospital; b) useful markers of airway inflammation/risk c) can identify people at with a higher likelihood of responding to anti-inflammatory therapy. The two tests we are mainly interested in are:

* Exhaled nitric oxide (measured with a portable handheld machine)
* The blood eosinophil count (obtained on a general blood test) +/- Other tests which we might be able to develop within this cohort (e.g. urine tests)

DETAILED DESCRIPTION:
BACKGROUND Asthma affects 10% of the general population but remains a diagnostic challenge. Considering the difficult access, weak specificity, and low clinical utility of bronchial provocation tests, more effective diagnostic methods are needed. Blood eosinophils and exhaled nitric oxide (FeNO) are biomarkers of type-2 inflammation that have established mechanistic, prognostic and theragnostic values in chronic asthma. Specifically, these biomarkers identify attack-prone patients with ongoing alarmin, type-2 cytokine, and chemokine signalling at the epithelial level driving airway hyperresponsiveness and accelerated lung function decline. Most importantly, these biomarkers also identify those who benefit the most from anti-inflammatory therapy. Considering the above clinical utilities, using biomarkers in primary care to diagnose airways disease in people with suspected asthma would represent a very effective diagnostic strategy.

HYPOTHESIS: In people with non-diagnostic spirometry and asthma suspected by primary care, measuring blood eosinophils and FeNO is a feasible diagnostic strategy with good accuracy and the added value of early mechanistic insight in epithelial signalling pathways.

OBJECTIVE: To estimate the diagnostic performance parameters of type-2 biomarkers in people with suspected asthma and a non-diagnostic spirometry. An exploratory analysis of inflammatory proteins (alarmin, type-2 cytokines, chemokines) in the nasal epithelial lining fluid (NELF) and serum according to biomarkers will be conducted. This and other secondary exploratory objectives will lead to better mechanistic and operational insight on the value of type-2 biomarkers in early disease.

METHODS: The investigators propose a prospective observational study on the logistical feasibility, receiver operating characteristics (ROC), and mechanistic value of point-of-care type-2 inflammatory biomarkers to diagnose asthma (Figure). The study will include 123 people ≥18 years old with non-diagnostic pre-postbronchodilator spirometry referred by primary care for a methacholine challenge via the Suspected Asthma pathway of the Centre Hospitalier Universitaire de Sherbrooke. After the methacholine challenge, patients will complete questionnaires, have blood eosinophils measured (by venous blood sample), FeNO measured (by electroluminescence), nasosorption performed, and serum harvested for allergy testing and inflammatory protein measurement.

OUTCOMES: The main analysis will be ROC plots of (1) FeNO alone; (2) blood eosinophils alone; and (3) the combination of blood eosinophils and FeNO;. The ROC plot will be based on a methacholine provocative dose ≤200 mcg (~ provocative concentration ≤8 mg/mL). The target sample size of 123 will have 90% power to compute 3 ROC curves' area under the curve (AUC) ≥ 0.7 significantly different from the null hypothesis (AUC=0.5) with a conservatively corrected two-sided α error < 0.016, assuming a positive/negative case ratio of 2. Secondary outcomes are the diagnostic and cost-effectiveness of blood eosinophil and FeNO measurement compared to methacholine challenges; and univariate plus multivariate modelling between blood eosinophils, FeNO, and inflammatory proteins (alarmins TSLP and IL-33; type-2 cytokines IL-4, -5, -13; chemokines eotaxin-3 and TARC) measured in the NELF and serum, or metabolites measured in the urine.

EXPECTED RESULTS: It is expected that type-2 inflammometry to be a useful alternative diagnostic pathway with benefits extending beyond diagnostic accuracy thanks to early insight into the inflammatory phenotype.

IMPACT: This observational study will support further validation studies and/or trials assessing biomarker-assisted diagnosis and management of asthma in the community setting. Measuring biomarkers at the time of diagnosis could facilitate a 'predict and prevent' approach to diagnostic algorithms in airway disease

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 12 years who have symptoms suggestive of asthma,
* referred by their primary care provider (defined as a non-respirologist, non-allergist, non-otolaryngologist) using the CHUS suspected asthma decision-making algorithm. Under that algorithm, patients have non-diagnostic pre- and post-bronchodilator spirometry and no contraindications to a methacholine challenge.
* Free and informed consent must be given by the patient (and their legal guardian, if applicable).

Exclusion Criteria:

* Use of an inhaled or systemic corticosteroid in the previous 48 hours;
* Smoking in the previous 6 hours; history of viral and/or bacterial respiratory infection in the past 4 weeks;
* major cardiopulmonary disease, including: a) chronic obstructive pulmonary disease (COPD), defined by all of the following: i) aged ≥ 40 years , ii) permanent obstruction on spirometry (FEV1/FVC <0.7) and iii) a smoking history of >10 pack-years or known alpha-1-antitrypsin deficiency, b) lung conditions deemed significant by the investigator, including cystic fibrosis and bronchiectasis, and c) unstable heart disease.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study has a collaboration agreement with the respiratory physiology service. In this context, a research invitation letter will be sent with confirmation of the appointment. The letter indicates that participation is voluntary and provides the expected length of the appointment (20-30 minutes), a QR code referring them to an online version of the Information and Consent Form (ICF), and a cell phone number and email address for the research team, with a phone number for individuals to state their refusal to be contacted. In the week preceeding the challenge, the clinical inhalation therapist will call non-objecting pre-screened patients to discuss the project and plan the study visit.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
AUC of the ROC analysis to diagnose asthma | FeNO measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg
Blood eosinophil count: ROC analysis AUC to diagnose asthma | Blood eosinophils measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg
Combination of FeNO + Blood eosinophil count: ROC analysis AUC to diagnose asthma | FeNO and blood eosinophils measured on the day of the methacholine challenge (i.e. Baseline visit)
  Diagnosis of asthma defined as a methacholine PD20 < 200 mcg

SECONDARY OUTCOMES:
Univariate association between biomarkers (blood eosinophils and FeNO) and inflammatory proteins/metabolites | Baseline
  Inflammatory proteins/metabolites measured in the NELF, serum, and urine. Further exploratory multivariate modelling adjusting for atopy (defined as a history of eczema, rhinoconjunctivitis, or food allergy and/or at least one sensitisation to an airbourne sensitiser) and biological sex.
Operational efficacy of the use of biomarkers as a diagnostic tool: | Baseline
  1. Potential reduction in diagnostic delay in asthma patients: the difference (in days) between the date of the challenge test and the date of the request
  2. Time difference (in minutes/days) for diagnosing asthma using biomarkers (FeNO + eosinophilia) versus a methacholine challenge.
  3. Cost difference between the use of biomarkers (traditional or point-of-care analysed separately) as 2nd diagnosis step versus a standard methacholine challenge test.
Biomarker level in asthmatic patients at time of diagnosis | Baseline
  Expressed as n (%) of diagnosed patients per square in a 3×3 grid stratified by combination of biomarkers (eosinophils <0.15, 0.015-<0.30, ≥0.30×109/L; FeNO <25, 25-<50, ≥50 ppb)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gronnier M, Desy L, Pouliot L, Lemieux SE, Vezina FA, Lachapelle P, Counil FP, Duval M, Cliche D, Lemaire-Paquette S, Coulibaly L, Hudon C, Lands LC, Ducharme FM, Tse S, Couillard S. Integrating blood eosinophils and exhaled nitric oxide (FeNO) in asthma diagnostic pathways for adults and children: the PROPULSION SANTE observational study with translational sub-studies (DIVE, DIVE2)-protocols. BMJ Open Respir Res. 2025 Nov 27;12(1):e003750. doi: 10.1136/bmjresp-2025-003750. PMID 41314665